CLINICAL TRIAL: NCT04837040
Title: A Randomized, Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Paltusotine in Subjects With Acromegaly Treated With Long-acting Somatostatin Receptor Ligands (PATHFNDR-1)
Brief Title: A Study to Evaluate the Safety and Efficacy of Paltusotine for the Treatment of Acromegaly
Acronym: PATHFNDR-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRN00808-09; 2020-005431-70 (EudraCT Number); 2024-511925-71-00 (EU CTIS Number)
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; PATHFNDR; Paltusotine; CRN00808
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paltusotine (Experimental)
  Interventions: Drug: Paltusotine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paltusotine — Paltusotine, tablets, once daily by mouth
  Other Names: CRN00808
  Arms: Paltusotine
Drug: Placebo — Placebo, tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled study designed to evaluate the safety and efficacy of paltusotine (also known as CRN00808; an orally administered nonpeptide somatostatin agonist) in subjects with acromegaly previously treated with somatostatin receptor ligand (SRL) based treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 years of age
2. Confirmed diagnosis of acromegaly and controlled (as measured by IGF-1 ≤1.0×ULN) via stable dose of protocol defined somatostatin receptor ligand therapy
3. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, or using effective method(s) of birth control
4. Willing to provide signed informed consent

Exclusion Criteria:

1. Treatment naïve or treatment-withdrawn acromegaly subjects
2. Prior treatment with paltusotine
3. Pituitary surgery within 24 weeks prior to Screening or history of pituitary radiation therapy
4. History or presence of malignancy except adequately treated basal cell and squamous cell carcinomas of the skin within the past 5 years
5. Use of any investigational drug within the past 30 days or 5 half-lives, whichever is longer
6. Known history of HIV, hepatitis B, or active hepatitis C
7. History of alcohol or substance abuse in the past 12 months
8. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this study
9. Cardiovascular conditions or medications associated with prolonged QT or those which predispose subjects to heart rhythm abnormalities
10. Subjects with symptomatic cholelithiasis
11. Subjects with clinically significant abnormal findings during the Screening Period, or any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the subject's safety or ability to complete the study
12. Subjects currently taking pasireotide LAR (within 24 weeks prior to Screening) or pegvisomant, dopamine agonists (within 12 weeks prior to Screening), or short acting somatostatin analogs (within 12 weeks prior to first dose of study drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2027-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (7):
  - Crinetics Study Site, Los Angeles, California
  - Crinetics Study Site, Torrance, California
  - Crinetics Study Site, Baltimore, Maryland
  - Crinetics Study Site, Boston, Massachusetts
  - Crinetics Study Site, Philadelphia, Pennsylvania
  - Crinetics Study Site, Pittsburgh, Pennsylvania
  - Crinetics Study Site, Nashville, Tennessee
- Argentina (3):
  - Crinetics Study Site, CABA, Buenos Aires
  - Crinetics Study Site, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Crinetics Study Site, Córdoba
- Crinetics Study Site, Ghent, Belgium
- Brazil (4):
  - Crinetics Study Site, Fortaleza, Ceará
  - Crinetics Study Site, Curitiba, Paraná
  - Crinetics Study Site, Porto Alegre, Rio Grande do Sul
  - Crinetics Study Site, Rio de Janeiro
- Crinetics Study Site, Sofia, Bulgaria
- France (2):
  - Crinetics Study Site, Bron
  - Crinetics Study Site, Pessac
- Hungary (2):
  - Crinetics Study Site, Budapest
  - Crinetics Study Site, Pécs
- Israel (2):
  - Crinetics Study Site, Beersheba
  - Crinetics Study Site, Petah Tikva
- Crinetics Study Site, Roma, Italy
- Crinetics Study Site, San Isidro, Lima region, Peru
- Poland (2):
  - Crinetics Study Site, Bydgoszcz
  - Crinetics Study Site, Poznan
- Russia (5):
  - Crinetics Study Site, Kemerovo, Kemerovo Oblast
  - Crinetics Study Site, Novosibirsk, Novosibirsk Oblast
  - Crinetics Study Site, Samara, Samara Oblast
  - Crinetics Study Site, Kazan', Tatarstan Republic
  - Crinetics Study Site, Moscow
- Crinetics Study Site, Belgrade, Serbia
- United Kingdom (3):
  - Crinetics Study Site, Sheffield, South Yorkshire
  - Crinetics Study Site, Coventry, West Midlands
  - Crinetics Study Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase 3, multicenter, randomized, placebo-controlled study where a total of 115 participants were screened, of which 58 participants were randomized (30 participants in the total paltusotine group and 28 participants in the placebo group) to the randomized control (RC) Phase.
Pre-assignment Details: Participants were randomized to treatment or placebo in a 1:1 ratio. Participants who completed the RC phase or who met rescue criteria could enter the open-label extension (OLE) phase. The RC Phase is completed. The OLE Phase is ongoing.
Groups:
- Paltusotine: Participants were randomized in a 1:1 ratio and received a daily dose paltusotine orally.
- Placebo: Participants were randomized to receive matching placebo tablets in a 1:1 ratio.
Period: RC Phase (Up to Week 36)
Arm/Group | Paltusotine | Placebo
Started | 30 | 28
Completed | 30 | 27
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: OLE Phase (Up to Week 240)
Arm/Group | Paltusotine | Placebo
Started | 27 | 26
Ongoing (OLE is ongoing) | 27 | 26
Completed | 0 | 0
Not Completed | 27 | 26

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined from the intention-to-treat principle and included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paltusotine | Placebo | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (14.57) | 53.9 (12.89) | 54.9 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 19
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 19 | 42
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintain Biochemical Response in IGF-1 (≤1.0× the Upper Limit of Normal [ULN]) at the End of the Randomized Control Phase (EOR)
Description: A value >1.0 indicates IGF-1 levels above the age- and sex-adjusted ULN. Response is defined as an IGF-1 level ≤1.0×ULN based on the average of last 2 measurements (weeks 34 and 36).
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- Paltusotine: Participants were randomized in a 1:1 ratio (paltusotine vs placebo) and received a daily dose paltusotine orally.
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 30 | 28
percentage of participants | 83.3 | 3.6
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Treatment comparison of all participants receiving paltusotine versus placebo has been presented; Test type: Superiority; p < 0.0001, exact logistic regression model; Odds Ratio (OR) = 126.526, 95% CI 2-sided [13.733 to 999.999]

2. Secondary Outcome: Change From Baseline in IGF-1 to EOR
Description: A value >1.0 indicates IGF-1 levels above the age- and sex-adjusted ULN. Baseline was defined as the last non-missing assessment prior to first dose of study drug for all assessments except IGF-1, growth hormone (GH), and acromegaly symptoms diary (ASD). Change from Baseline was determined by calculating (post-Baseline value - Baseline value).
Time Frame: Baseline to 36 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: nanograms per milliliter (ng/ml)
Groups:
- Paltusotine: Participants were randomized in a 1:1 ratio and received a daily dose of paltusotine orally.
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 30 | 28
nanograms per milliliter (ng/ml) | 0.042 (0.0932) | 0.833 (0.0962)
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; least squares means difference = -0.791, 95% CI 2-sided [-1.057 to -0.525]

3. Secondary Outcome: Percentage of Participants With GH <1.0 ng/mL at Week 34
Description: GH maintenance of response was analyzed in participants with GH<1.0 ng/mL at week 34, out of those who had GH<1.0 ng/mL at Baseline, using the same methodology as the primary endpoint.
Time Frame: Week 34
Population: Full Analysis Set. Only those participants with data available at specified timepoints have been presented.
Measure: Number; unit: percentage of participants
Groups:
- Paltusotine: Participants were randomized in a 1:1 ratio (paltusotine vs placebo) and received a daily dose of paltusotine orally.
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 23 | 18
percentage of participants | 87.0 | 27.8
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Treatment comparison of all participants receiving paltusotine versus placebo has been presented; Test type: Superiority; p = 0.0003, exact logistic regression model; Odds Ratio (OR) = 16.609, 95% CI 2-sided [2.864 to 181.355]

4. Secondary Outcome: Change From Baseline in Total Acromegaly Symptoms Diary (ASD) Score to EOR
Description: The ASD is a sponsor-developed daily diary to assess important acromegaly symptoms from the patient perspective. The weekly average ASD total score is calculated from 7 items associated with acromegaly (headache pain, joint pain, sweating, fatigue, weakness in legs, swelling, and numbness or tingling). The ASD total score ranges from 0 to 70 with each symptom contributing up to 10 points. A higher score = higher symptom severity. Change from baseline in total ASD was defined as the postbaseline total ASD score (the average of the available scores seven days on or prior to the scheduled visit date) minus the baseline total ASD score.
Time Frame: Baseline to 36 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 30 | 28
units on a scale | -0.606 (1.5044) | 4.558 (1.5926)
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Test type: Superiority; p = 0.0216, ANCOVA; least square mean difference = -5.164, 95% CI 2-sided [-9.536 to -0.792]

ADVERSE EVENTS:
Time Frame: Up to 36 Weeks
Description: Serious TEAEs and TEAEs were collected in a safety analysis set which was comprised of all participants who received study drug with treatment assignment based on the treatment received. The adverse events are presented as of last participant visit in the RC phase only. Final adverse events from the ongoing OLE will be reported after study completion. All participants, irrespective of their dose level in the paltusotine or placebo arms, have been presented.
Arm/Group | Paltusotine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/28
Other Adverse Events (participants affected / at risk) | 24/30 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paltusotine (N=30) | Placebo (N=28)
cholecystitis acute (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paltusotine (N=30) | Placebo (N=28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Peripheral swelling (General disorders) | 2 | 10
Fatigue (General disorders) | 2 | 5
Asthenia (General disorders) | 1 | 4
Hyperhidrosis (General disorders) | 0 | 4
Headache (Nervous system disorders) | 6 | 10
Paraesthesia (Nervous system disorders) | 0 | 7
Dizziness (Nervous system disorders) | 1 | 2
COVID-19 (Infections and infestations) | 0 | 6
Urinary tract infection (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT04837040/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT04837040/SAP_001.pdf